CLINICAL TRIAL: NCT00666328
Title: The Evaluation of Patients With Acute Hypertension and Intracerebral Hemorrhage With Intravenous Clevidipine Treatment (ACCELERATE)
Brief Title: Clevidipine in the Treatment of Patients With Acute Hypertension and Intracerebral Hemorrhage (ACCELERATE)
Acronym: ACCELERATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-07-02
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension; Hemorrhage
Keywords: Hypertension; Hemorrhage; Intracranial Pressure; Antihypertensive Agent; Calcium Channel Blocker
MeSH Terms: conditions — Hypertension; Hemorrhage | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clevidipine (Experimental): This will be a single-arm study with no reference therapy.
  Interventions: Drug: clevidipine

INTERVENTIONS:
Drug: clevidipine — Clevidipine injectable emulsion (0.5 mg/mL) in 20% lipid emulsion in 100 mL bottles was administered intravenously to all patients via a single dedicated line.
  Clevidipine was infused at an initial rate of 2.0 mg/h for the first 1.5 minutes. Thereafter, titration to higher infusion rates were to be attempted as needed to obtain the target systolic blood pressure (SBP) range (SBP ≤160 mmHg to ≥140 mmHg). Titration to effect was to proceed by doubling the dose every 1.5 minutes, up to a maximum of 32.0 mg/h, until the desired effect (SBP within the target range) was attained. The clevidipine infusion rate could be increased or decreased to maintain systolic blood pressure for up to a maximum of 96 hours.
  Other Names: clevidipine injectable emulsion; clevidipine emulsion; Cleviprex

SUMMARY:
The purpose of this study was to determine the efficacy and safety of clevidipine for treating acute hypertension (high blood pressure, defined as systolic blood pressure >160 mmHg) in patients with intracerebral hemorrhage (i.e., bleeding in the brain; stroke).

DETAILED DESCRIPTION:
This was a multicenter, single-arm, non-blinded dose titration efficacy and safety trial evaluating the ability of clevidipine, a vascular-selective L-type calcium channel antagonist, to rapidly control acute hypertension in patients with intracerebral hemorrhage. Informed consent was obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures. At screening, a clinical and neurological examination was carried out. For the purposes of this study, acute hypertension was defined as SBP >160 mmHg immediately prior to initiation of study drug. Approximately 30 to 40 patients with acute intracerebral hemorrhage (ICH) were planned to be enrolled with approximately 10 patients requiring monitoring of intracranial pressure (ICP). Infusion of study drug was initiated within 12 hours of ICH symptom onset. All eligible patients enrolled received clevidipine in an open label manner. Clevidipine was to be infused at an initial rate of 2.0 mg/h for the first 1.5 minutes. Thereafter, titration to higher infusion rates were to be attempted as needed, to obtain the target SBP range (SBP ≤160 mmHg to ≥140 mmHg). Titration to effect was to proceed by doubling the dose every 1.5 minutes, up to a maximum of 32.0 mg/h, until the desired effect (SBP within the target range) was attained. During the first 30 minutes, if the desired blood pressure lowering effect was not attained or maintained, an alternative intravenous (IV) antihypertensive agent(s), advised to be a different class other than calcium channel blockers, could be used with or without stopping the clevidipine infusion. The clevidipine infusion could continue for up to a maximum of 96 hours. Twenty-four hour follow-up computerized tomography (CT) scan results were recorded, including measurement of intracerebral hematoma volumes. Assessment of safety was performed throughout the treatment period and until 6 hours after termination of study drug. Patients were followed for 7 days following termination of the clevidipine infusion.

ELIGIBILITY:
Inclusion Criteria:

* CT evidence of intracerebral hemorrhage (diagnosis and treatment within 12 hours of symptom onset)
* Age 18 years or older
* Baseline systolic blood pressure (immediately prior to initiation of clevidipine) >160 mmHg measured using an arterial line. ICP-monitored patients enrolled in the sub-study were enrolled if SBP at the time of enrollment was ≤160 mmHg
* Required antihypertensive therapy to achieve systolic blood pressure ≤160 mmHg
* Written informed consent obtained

Exclusion Criteria:

* Decision for early surgical evacuation prior to 30 minutes of clevidipine
* Receipt of an oral antihypertensive within 2 hours prior to initiation of clevidipine
* Treatment with a continuous infusion of an IV antihypertension agent prior to initiation of clevidipine. Bolus treatment with urapidil (Germany only), labetalol or hydralazine was permitted. ICP-monitored patients enrolled in the sub-study could be enrolled with a continuous infusion of an IV antihypertensive agent prior to the initiation of clevidipine.
* Intracerebral hematoma considered to be related to trauma by the neurologist or neurosurgeon
* Aneurysmal sub-arachnoid hemorrhage
* Glasgow coma score of <5 and fixed dilated pupils
* Expectation that the patient would not tolerate or require intravenous antihypertensive therapy for a minimum of 30 minutes
* Known or suspected aortic dissection
* Acute myocardial infarction on presentation
* Positive pregnancy test or known pregnancy
* Intolerance or allergy to calcium channel blockers
* Allergy to soybean oil or egg lecithin
* Known liver failure, cirrhosis or pancreatitis
* Prior directives against advanced life support
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Graffagnino, MD, Principal Investigator — Duke University
Locations (17):
- United States (14):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - The Queens Medical Center, Honolulu, Hawaii
  - The John Hopkins Hospital, Baltimore, Maryland
  - Maine Medical Center, Portland, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Guilford Neurologic - Moses H Cone Health System, Greensboro, North Carolina
  - Cleveland Clinic Hospitals, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University Stroke Research, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University Health Science Center at S.A., San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
- Germany (3):
  - Universitätsklinikum Leipzig, Liebigstraße 22a, Leipzig
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Heidelberg, Heidelberg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients considered for inclusion in this study were recruited from June 2008 through April 2010 primarily from hospital emergency departments and Neurology Intensive Care Units, having presented with acute hypertension and intracerebral hemorrhage (ICH). Enrollment targeted a subset of ~10 patients requiring intracranial pressure (ICP) monitoring.
Pre-assignment Details: Participants were required to have a systolic blood pressure (SBP) greater than 160 mm Hg both prior to enrollment and immediately prior to study drug initiation. Participants with SBP </=160 mm Hg immediately prior to study drug did not receive clevidipine and were treated per standard of care.
Groups:
- Clevidipine: Clevidipine was administered to eligible participants via intravenous infusion at a starting dose of 2.0 mg/h for 1.5 minutes. Clevidipine was titrated to effect thereafter by doubling the dose every 1.5 minutes, as tolerated by the patient, up to a maximum dose of 32 mg/h, to lower blood pressure within the protocol specific target range (SBP ≤160 mmHg to ≥140 mmHg) for a minimum of 30 minutes and up to 96 hours.
Period: Overall Study
Arm/Group | Clevidipine
Started | 35 (Safety population: participants dosed with study drug (primary population for Safety analyses))
Modified Intent To Treat (mITT) | 33 (mITT population: participants dosed and in whom all inclusion and no exclusion criteria were met)
Completed | 30 (30/35 completed the study within the Safety population; 28/33 completed within the mITT population.)
Not Completed | 5
Not completed — Death | 2
Not completed — Lost to Follow-up | 2
Not completed — No longer met eligibility criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- Clevidipine: mITT (Modified Intent To Treat) Population (n=33): This population is the primary population for the efficacy analyses.
  Clevidipine was administered to eligible participants via intravenous infusion at a starting dose of 2.0 mg/h for 1.5 minutes. Clevidipine was titrated to effect thereafter by doubling the dose every 1.5 minutes, as tolerated by the patient, up to a maximum dose of 32 mg/h, to lower blood pressure within the protocol specific target range (SBP ≤160 mmHg to ≥140 mmHg) for a minimum of 30 minutes and up to 96 hours. Clevidipine was titrated up or down as necessary to maintain blood pressure within the target range.
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: participants] | 63.9 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0
  Asian | 3
  Black or African American | 9
  Native Hawaiian or Pacific Islander | 0
  White | 21
Baseline Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 186.5 (20.39)
Baseline Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 85.7 (12.89)

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Achieve Target SBP Range (≤160 mmHg to ≥140 mmHg) Within 30 Minutes of Initiation of Clevidipine
Description: The median time, in minutes, was estimated with its two-tailed 95% confidence interval from the time of the initiation of clevidipine infusion until the first observed SBP was achieved in the target range of ≤160 mmHg to ≥140 mmHg within the first 30 minutes of clevidipine treatment. If patients did not reach the blood pressure target range within the first 30 minutes, their data was considered censored at 30 minutes. If another IV and/or oral antihypertensive agent indicated for hypertension was administered less than 30 minutes prior to achieving the endpoint, the data was considered censored at the time when the additional or alternative antihypertensive agent was given.
Time Frame: Within 30 minutes of study drug initiation
Population: Modified Intent To Treat (mITT) population: all participants dosed with clevidipine and in whom all inclusion criteria and none of the exclusion criteria were met.
Measure: Median (95% Confidence Interval); unit: minutes
Groups:
- Clevidipine: Clevidipine was administered via intravenous infusion at a starting dose of 2.0 mg/h for 1.5 minutes and titrated to effect thereafter by doubling the dose every 1.5 minutes, as tolerated by the patient, up to a maximum dose of 32 mg/h, to lower blood pressure within the protocol specific target range (SBP ≤160 mmHg to ≥140 mmHg). Clevidipine was titrated up or down, as necessary, to maintain blood pressure within the target range for a minimum of 30 minutes to a maximum of 96 hours.
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
minutes | 5.5 [3 to 10]

2. Secondary Outcome: Percentage of Participants Achieving a SBP of ≤160 mmHg Within 30 Minutes of Initiation of Clevidipine
Description: The percentage of patients who reached SBP of ≤160 mmHg within the first 30 minutes of initiation of clevidipine infusion was summarized. If an additional or alternative IV antihypertensive agent and/or oral antihypertensive agent was administered for hypertension prior to a patient achieving SBP≤160 mmHg during the initial 30-minute treatment period, then the patient was considered to have failed to reach this efficacy endpoint.
Time Frame: Within 30 minutes of study drug initiation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
percent participants | 97 [84.2 to 99.9]

3. Secondary Outcome: Percent Change From Baseline in Systolic Blood Pressure During the Initial 30 Minutes of Clevidipine Infusion
Description: Over the initial 30 minutes of the treatment period, the percent change from baseline (defined as immediately prior to study drug initiation) was summarized descriptively at 1, 2, 3, 4, 5, 6, 7, 10, 15, 20, 25, and 30 minutes after clevidipine initiation. Decreases in SBP from baseline were observed over the course of this time period.
Time Frame: Baseline through 30 minutes post initiation of clevidipine infusion
Measure: Mean (Standard Deviation); unit: percent change in SBP
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
percent change in SBP
  Baseline Through Initial 1 Min. | -2.2 (5.76)
  Baseline Through Initial 2 Min. | -4.7 (9.43)
  Baseline Through Initial 3 Min. | -5.9 (8.95)
  Baseline Through Initial 4 Min. | -8.5 (8.54)
  Baseline Through Initial 5 Min. | -9.8 (9.15)
  Baseline Through Initial 6 Min. | -11.3 (10.54)
  Baseline Through Initial 7 Min. | -13.9 (9.92)
  Baseline Through Initial 10 Min. | -14.0 (11.52)
  Baseline Through Initial 15 Min. | -17.4 (12.20)
  Baseline Through Initial 20 Min. | -17.4 (11.75)
  Baseline Through Initial 25 Min. | -18.9 (10.68)
  Baseline Through Initial 30 Min. | -20.0 (8.16)

4. Secondary Outcome: Magnitude, Frequency and Duration of Systolic Blood Pressure Excursions (Calculated as Area Under the Curve [AUC]) Outside the Target Range Normalized Per Hour for the Duration of the Clevidipine Monotherapy Infusion
Description: Total AUC-SBP captures the magnitude and duration of SBP either above the upper limit of the target SBP range at 160 mm Hg or below the lower limit of 140 mm Hg and normalized per hour for the duration of clevidipine infusion. A larger value for AUC-SBP indicates greater SBP variability outside the target range.
Time Frame: Duration of the study drug infusion (up to 96 hours)
Measure: Mean (Standard Deviation); unit: mm Hg × min/hr
Groups:
- Clevidipine: Clevidipine was administered via intravenous infusion at a starting dose of 2.0 mg/h for 1.5 minutes and titrated to effect thereafter by doubling the dose every 1.5 minutes, as tolerated by the patient, up to a maximum dose of 32 mg/h to lower blood pressure within the protocol specific target range (SBP ≤160 mmHg to ≥140 mmHg) for 30 minutes to 96 hours. Clevidipine was titrated up or down as necessary to maintain blood pressure within the target range.
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
mm Hg × min/hr | 347.7 (323.06)

5. Secondary Outcome: Percent Time Blood Pressures Were Maintained Within the Target Range (Systolic Blood Pressure ≤160 mmHg to ≥140 mmHg) Over Each 24 Hour Period During Monotherapy Infusion of Clevidipine
Description: The percent time that SBP was maintained within the SBP target range (≤160 mmHg to ≥140 mmHg) was summarized for each 24-hour period of monotherapy of clevidipine infusion through 96 hours (0 -≤24 h, 24-≤48 h, 48-≤72 h, 72-≤96 h). For purposes of this analysis, SBP data were available from all mITT patients for the overall infusion period and from 0 to ≤24 hours of infusion; however, data was only available for 8 patients from 24 to ≤48 hours, 4 patients from 48 to ≤72 hours and 1 patient from 72 to ≤96 hours due to the variability in infusion durations >24 hours across patients.
Time Frame: From study drug initiation through termination (up to 96 h)
Population: The Modified Intent-to-Treat (mITT) population, defined as all enrolled patients who are eligible for the study (i.e., meet all the inclusion criteria and do not meet any of the exclusion criteria) and treated with clevidipine infusion, population will be the primary population for the efficacy analyses.
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
percent time
  0 -≤24 h of clevidipine infusion; n=33 | 51.91 (25.46)
  24-≤48 h of clevidipine infusion; n=8 | 61.12 (21.14)
  48-≤72 h of clevidipine infusion; n=4 | 46.94 (33.25)
  72-≤96 h of clevidipine infusion; n=1 | 65.91 (0.00)

6. Secondary Outcome: Mean Dose of Clevidipine During the Treatment Period
Description: Mean total dose of clevidipine from study drug initiation to the end of clevidipine treatment
Time Frame: Up to 96 hours
Population: The Safety population is defined as all enrolled patients who are dosed with clevidipine. This population serves as the primary population for the safety analyses.
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Clevidipine
Number analyzed (Participants) | 35
milligrams (mg) | 260.28 (321.68)

7. Secondary Outcome: Median Dose of Clevidipine During the Treatment Period
Description: Mean total dose of clevidipine from study drug initiation to the end of clevidipine treatment
Time Frame: Up to 96 hours
Measure: Median (Inter-Quartile Range); unit: milligrams (mg)
Arm/Group | Clevidipine
Number analyzed (Participants) | 35
milligrams (mg) | 116.32 [0.7 to 1213.8]

8. Secondary Outcome: Proportion of Patients Requiring an Additional or Alternative Antihypertensive Agent(s) With or Without Clevidipine
Description: Additional or alternative antihypertensive agent(s) comprise the use of other antihypertensive agent(s) either with clevidipine (additional) or in place of clevidipine (alternative) for the indication of hypertension from the time of clevidipine initiation to clevidipine termination. For purposes of this analysis, additional or alternative antihypertensive agents did not include oral antihypertensives that were administered in order to transition IV clevidipine-treated patients to oral therapy during the transition period of the study.
Time Frame: Up to 96 hours
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 33
participants | 18

9. Secondary Outcome: Percent Change in Heart Rate During 30 of Initiation of Clevidipine
Description: Multiple timepoints were assessed (minutes 1, 2, 3, 4, 5, 10, 15, 20, 30) for analysis of percent change in heart rate during the initial 30 minutes.
Time Frame: From study drug initiation through each specified timepoint
Population: The Safety population is defined as all enrolled patients who are dosed with clevidipine. This population serves as the primary population for the safety analyses. Data for 33 of the 35 patients in the Safety population had data for the 30 minute time point used for this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Clevidipine
Number analyzed (Participants) | 35
percent change
  Study Drug Initiation Through Initial 1 Min; n=35 | -0.4 (5.02)
  Study Drug Initiation Through Initial 2 Min; n=32 | -0.7 (5.30)
  Study Drug Initiation Through Initial 3 Min; n=35 | -0.3 (6.41)
  Study Drug Initiation Through Initial 4 Min; n=34 | 0.2 (8.22)
  Study Drug Initiation Through Initial 5 Min; n=34 | 2.1 (8.25)
  Study Drug Initiation Through Initial 6 Min; n=34 | 2.6 (7.73)
  Study Drug Initiation Through Initial 7 Min; n=34 | 2.5 (9.30)
  Study Drug Initiation Through Initial 10 Min; n=34 | 5.6 (13.67)
  Study Drug Initiation Through Initial 15 Min; n=35 | 5.5 (15.65)
  Study Drug Initiation Through Initial 20 Min, n=35 | 6.2 (15.44)
  Study Drug Initiation Through Initial 25 Min; n=35 | 5.4 (14.50)
  Baseline Through Initial 30 Mins; n=33 | 4.9 (14.41)

10. Secondary Outcome: The Percentage of Patients Whose Systolic Blood Pressure is <90 mmHg Within 30 Minutes of the Initiation of Clevidipine Infusion
Time Frame: Within 30 minutes of the initiation of study drug infusion
Population: as for outcome 6
Measure: Number; unit: percent participants
Arm/Group | Clevidipine
Number analyzed (Participants) | 35
percent participants | 0

ADVERSE EVENTS:
Time Frame: AEs occurring from initiation of clevidipine infusion until up to 6 hours after cessation of clevidipine and SAEs that occurred from initiation of clevidipine infusion until up to 7 days after cessation of clevidipine infusion were assessed.
Groups:
- Clevidipine: Safety Population (n=35): This population is the primary population for the safety analyses.
  Clevidipine was administered to eligible participants via intravenous infusion at a starting dose of 2.0 mg/h for 1.5 minutes. Clevidipine was titrated to effect thereafter by doubling the dose every 1.5 minutes, as tolerated by the patient, up to a maximum dose of 32 mg/h, to lower blood pressure within the protocol specific target range (SBP ≤160 mmHg to ≥140 mmHg) for a minimum of 30 minutes and up to 96 hours. Clevidipine was titrated up or down as necessary to maintain blood pressure within the target range.
Arm/Group | Clevidipine
Serious Adverse Events (participants affected / at risk) | 9/35
Other Adverse Events (participants affected / at risk) | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clevidipine (N=35)
Cardio-respiratory arrest (Cardiac disorders) | 1 — unrelated
Supraventricular tachycardia (Cardiac disorders) | 1 — unrelated
Brain oedema (Nervous system disorders) | 2 — unlikely related
Cerebral haematoma (Nervous system disorders) | 1 — unrelated
Convulsion (Nervous system disorders) | 1 — unlikely related
Haemorrhage intracranial (Nervous system disorders) | 1 — unlikely related
Intraventricular haemorrhage (Nervous system disorders) | 1 — unrelated
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — unrelated
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clevidipine (N=35)
Hypotension (Vascular disorders) | 3 — 1 patient (2.86%) discontinued study drug due to a TEAE of hypotension(baseline SBP 82/47 mm Hg). This was a non-serious AE moderate in severity and related to study treatment. The AE lasted 51 min and resolved 29 minutes after study drug withdrawal.
Leukocytosis (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomitting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 7
Blood creatinine increased (Investigations) | 2
Prothrombin time prolonged (Investigations) | 2
White blood cell count increased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyposphataemia (Metabolism and nutrition disorders) | 4
Headache (Nervous system disorders) | 5
Agitation (Psychiatric disorders) | 4
Urinary retention (Renal and urinary disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site agrees that it will not publish until the earlier of presentation and publication of results or until 12 months after study conclusion. The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 90 days from the time submitted to the sponsor for review in order to allow sponsor time to file any patent applications. The sponsor cannot require changes to the communication and cannot extend the embargo.